CLINICAL TRIAL: NCT05941247
Title: A Phase I, Single-arm, Open-label, Ethnobridging Study to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) of Single and Multiple Oral Doses of Hemay005 Tablets in Healthy Caucasian Adult Volunteers
Brief Title: A Study to Evaluate the Effects of Single and Multiple Doses of Hemay005 Tablets in Health Caucasian Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ganzhou Hemay Pharmaceutical Co., Ltd (Industry)
Collaborators: Hemay Pharmaceutical PTY. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HM005PS1S05
Record Dates: First submitted 2023-04-05; First posted 2023-07-12 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: PK parameters; Caucasian
MeSH Terms: interventions — Hemay005

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemay005 60 mg (Experimental): The participant will receive single administration of Hemay005 tablets at dose of 60 mg on Day 1. Thereafter, those participants will receive Hemay005 tablets at dose of 60 mg for 7 consecutive days, which will be administrated twice daily.
  Interventions: Drug: Hemay005 60 mg

INTERVENTIONS:
Drug: Hemay005 60 mg — The eligible healthy adult participants will enter Single-dose Administration Period, receiving a single administration of Hemay005 tablets orally at a dose of 60 mg on Day 1 morning under fasted condition.
  On Day 3, those participants will receive Hemay005 tablets at dose of 60 mg for 7 consecutive days, which will be administrated twice daily (BID) during Day 3 to Day 8 and only in the morning on Day 9.
  Other Names: Hemay005 treatment group

SUMMARY:
The purpose of the study is to assess the safety and tolerability of single and multiple oral doses of Hemay005 tablets in healthy Caucasian adult volunteers.

DETAILED DESCRIPTION:
This is a phase I, single-arm, open-label ethno-bridging study. The study is being conducted to test a potential new treatment for Behçet's disease (BD) called Hemay005.

The primary objective of this study is to evaluate the safety and tolerability of Hemay005 tablets after single and multiple oral doses in healthy Caucasian adult volunteers. The secondary objective of this study is to assess the pharmacokinetic parameters (time to remove the study drug from blood) of Hemay005 tablets after single and multiple oral doses.

The results of Chinese healthy volunteers will be used as a historical control to compare the ethnic differences between Chinese and Caucasians.

Approximately 12 eligible healthy (Caucasian) adult participants (male: female = 1:1) will be enrolled in this study.

The participant will be screened to determine their suitability to take part in the study within 28 days before receiving a dose of the study treatment. There will be one confinement period in the clinic, which will start on the day before dosing with dosing on Day 1 and discharge on Day 11. The participant will be asked to attend the clinic for a final study visit on Day 20. This visit will be the end of the participation in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female Caucasian participants (male: female = 1:1) between 18 and 55 years of age (both inclusive) at the time of signing the informed consent.
2. Body weight between 50 and 100 kg (both inclusive) for males or between 45 and 100 kg (both inclusive) for females; and body mass index (BMI) within 18-32 kg/m2 (both inclusive).
3. In good health as determined by screening tests. Good health is defined as having no clinically relevant abnormalities identified by a detailed medical history, full physical examination, vital signs (including measurement of body temperature, HR, blood pressure and respiratory rate), 12-lead ECG, and clinical laboratory tests.
4. Female participants must not be pregnant or breastfeeding and must use an effective contraception method from informed consent obtained to 180 days after last dose administration, with the exception of participants who have undergone sterilization in the preceding 3 months, or who are postmenopausal.

   A woman of childbearing potential (WOCBP) must undergo pregnancy testing prior to the first dose of the investigational medicinal product (IMP). The participant must be excluded from the study if the serum pregnancy test is positive. A postmenopausal state is defined as 12 months of amenorrhea without an alternative medical cause. In the absence of 12 months of amenorrhea, menopause may be confirmed by follicle-stimulating hormone (FSH) measurement. Females on hormonal replacement therapy (HRT), where menopausal status is indeterminate, will be required to use a non-estrogen hormonal contraceptive method if they wish to continue their HRT during the study. Participants must otherwise discontinue HRT to allow for confirmation of postmenopausal status prior to enrollment in the study.

   Males who are sexually active and who are partners of women of childbearing potential must agree to use an effective contraception from informed consent obtained to 180 days after last dose administration.
5. A negative result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
6. Provide written informed consent prior to undertaking any study-related procedures.
7. Must not be under any administrative or legal supervision or under institutionalization as per a regulatory or juridical order.

Exclusion Criteria:

1. Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, musculoskeletal, rheumatological, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
2. Any history or presence of gastrointestinal, hepatic, renal disease that affect drug absorption or metabolism.
3. Any history or presence of chronic infectious diseases such as tuberculosis (TB) (judged by the Investigator according to QuantiFERON-TB Gold).
4. Presence or history of drug/food hypersensitivity, or anaphylactic reaction, diagnosed and treated by a physician, or have special dietary requirements.
5. Known hypersensitivity to any component of the IMP formulation.
6. Any surgery within 1 months prior to the first dose.
7. Positive result on any of the following tests: hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), hepatitis B core antibodies (HBcAb) (for those with positive result on HbcAb, a HBV deoxyribonucleic acid (DNA) test will be performed and those with positive HBV DNA results will be excluded), HCV antibody (HCVAb), anti-human immunodeficiency virus 1 and 2 antibodies.
8. History or presence of alcohol abuse (defined as alcohol consumption more than 2 units per day 6 months prior to the first dose, 1 unit=360 mL of beer or 45 mL of alcohol 40% and above or 150 mL of wine).
9. History of drug abuse including narcotic and psychiatric drugs within 1 year prior to screening or a positive drug abuse test result at screening. One repeat is allowed at the discretion of the study doctor in case of false positives.
10. Regular smoking (defined as more than 5 cigarettes or equivalent per week) within one year prior to the first dose, or unable to stop smoking from 48 hours prior to the first drug administration to the last time point for collecting PK blood samples (Day 11).
11. Positive alcohol test at screening and check-in on Day -1.
12. Any consumption of xanthine bases and/or grapefruit or products containing xanthine bases and/or grapefruit within 2 weeks prior to the first dose; or unable to stop consumption of above ingredients during the pharmacokinetic (PK) assessments period (Day 1 to Day 11).
13. Any consumption of chocolate or caffeine or products containing caffeine within 48hours prior to the first dose; or unable to stop consumption of above ingredients during the PK assessments period (Day1 to Day11).
14. Any consumption of alcohol or products containing alcohol within 48 hours prior to study site admission (Day -1); or unable to stop consumption of alcohol during the PK assessments period (Day 1-Day 11).
15. Any drug that inhibits or induces liver drug metabolism (inducers include barbiturates, carbamazepine, rifampicin, phenytoin, glucocorticoids, omeprazole, etc.; inhibitors include selective serotonin reuptake inhibitor (SSRI) antidepressants, cimetidine, diltiazem, macrolides, nitroimidazoles, sedative-hypnotics, verapamil, fluoroquinolones, antihistamines, etc.) within 30 days prior to the first dose or during the study.
16. Any prescription medication, within 14 days prior to administration of the first dose, with the exception of hormonal contraception, menopausal hormone replacement therapy or occasional analgesics such as Paracetamol, Ibuprofen and standard daily vitamins etc. in short term at the Investigator's direction.
17. Made a blood donation of greater than 400 ml within 4 weeks prior to the first dose or during the study.
18. Any participant who enrolled in or participated in any other clinical study involving an investigational product, or in any other type of medical research within 1 month or within 5 times the elimination t1/2 prior to administration of the first dose.
19. Any vaccination in the 14 days prior to administration of the first dose.
20. Any participant who, in the judgment of the Investigator, is likely to be non-compliant during the study, or to be unable to cooperate due to language problems or poor mental development.
21. Any participant who is the Investigator, research assistant, pharmacist, study coordinator, or other staff thereof directly involved in conducting the study or any person dependent on (employees or immediate family members) the study site, the Investigator or the Sponsor.
22. Any participant who cannot be contacted in the case of an emergency.
23. Any participant in whom venous blood collection is difficult.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AE) following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  Incidence and severity of adverse events as assessed by CTCAE V5.0 by the investigator.
Number of participants with abnormal hematology laboratory tests results following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by Clinical laboratory abnormality in hematology assessed by changes from baseline following administration of Hemay005 tablets
Number of participants with abnormal chemistry laboratory tests results following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by Clinical laboratory abnormality in clinical chemistry assessed by changes from baseline following administration of Hemay005 tablets
Number of participants with abnormal coagulation laboratory tests results following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by Clinical laboratory abnormality in coagulation assessed by changes from baseline following administration of Hemay005 tablets
Number of participants with abnormal urinalysis results following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by Clinical laboratory abnormality in urinalysis assessed by changes from baseline following administration of Hemay005 tablets
Number of participants with abnormal stool analysis results following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by Clinical laboratory abnormality in stools assessed by changes from baseline following administration of Hemay005 tablets
Number of participants with abnormal systolic and diastolic blood pressure following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by changes in Vital signs from baseline measuring blood pressure. Blood pressure is measured by placing the stethoscope over the arm.
Number of participants with abnormal heart rate following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by changes in Vital signs from baseline measuring heart rate. Heart Rate is measured by an ECG and respiration rate is counted manually as breaths per minute by the Clinical Unit Assistants.
Number of participants with abnormal body temperature following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  The safety and tolerability of Hemay005 tablets will be assessed by changes in Vital signs from baseline measuring body temperature. Body temperature is measured using an oral thermometer.
Number of participants with abnormal electrocardiograms readings following administration of Hemay005 tablets as a measure of safety and tolerability | Up to Day 20 after the first dose
  12-lead ECGs will be obtained during the study using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT, and QT duration corrected for heart rate by Fridericia's formula (QTcF intervals) at each timepoint

SECONDARY OUTCOMES:
Change from baseline in the maximum plasma concentration (Cmax) following administration of Hemay005 tablets to evaluate the pharmacokinetics (PK) characteristics of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the maximum plasma concentration (Cmax)
Change from baseline in time to Cmax (Tmax) following administration of Hemay005 tablets to evaluate the pharmacokinetics (PK) characteristics of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the time to Cmax (Tmax)
Area under the curve from time 0 to the last measurable concentration (AUC0-t) to evaluate the Pharmacokinetic (PK) parameters of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the area under the curve from time 0 to the last measurable concentration (AUC0-t)
Area under the curve from time 0 extrapolated to infinite time (AUC0-inf) to assess the Pharmacokinetic (PK) parameters of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the area under the curve from time 0 extrapolated to infinite time (AUC0-inf),
Change from Baseline in half-life (t1/2) following administration of Hemay005 tablets to evaluate the pharmacokinetics (PK) characteristics of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the half-life (t1/2)
Change from Baseline in apparent clearance (CL/F) following administration of Hemay005 tablets to evaluate the pharmacokinetics (PK) characteristics of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the apparent clearance (CL/F)
Change from Baseline in apparent volume of distribution (Vz/F) following administration of Hemay005 tablets to evaluate the pharmacokinetics (PK) characteristics of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the apparent volume of distribution (Vz/F)
Change from Baseline in serum trough concentration (Ctrough) following administration of Hemay005 tablets to evaluate the pharmacokinetics (PK) characteristics of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the serum trough concentration (Ctrough)
Area under the curve extrapolated as a percentage of the total (AUC_%Extrap) to assess the Pharmacokinetic (PK) parameters of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring the area under the curve extrapolated as a percentage of the total (AUC_%Extrap)
Change from Baseline in mean residence time from the time of dosing to the time of last measurable concentration (MRTlast) to assess the Pharmacokinetic (PK) parameters of Hemay005 tablets | On Day 1 and Day 9, blood samples for PK analysis will be collected within 1 hour pre-dose, 0.5, 1, 1.5, 2, 3, 5, 8, 12, 16, 24, 36 and 48 hours post-dose; during Day 4 to Day 8 in the morning prior to administration.
  The PK parameters are assessed by measuring mean residence time from the time of dosing to the time of last measurable concentration (MRTlast)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Argent, Principal Investigator — Scientia Clinical Research Ltd
Locations (1):
- Scientia Clinical Research Ltd, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to other researchers.